CLINICAL TRIAL: NCT04826302
Title: Efficacy of Myofascial Induction as a Manual Therapy Technique in Patients With Anxiety. A Randomized Double Blind Clinical Trial Controlled With Placebo
Brief Title: Efficacy of Myofascial Induction as a Manual Therapy Technique in Patients With Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Complutense de Madrid (Other)
Responsible Party: Principal Investigator, Rodrigo Gozalo Pascual, Physical / Manual Therapist (PT, PhD Student), Biomechanics Professor, Universidad Complutense de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MyofascialAnxiety
Record Dates: First submitted 2021-03-25; First posted 2021-04-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Anxiety
Keywords: anxiety; myofascial induction; myofascial release; manual therapy; physiotherapy
MeSH Terms: conditions — Anxiety Disorders | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: A randomized double blind clinical trial controlled with placebo in which neither the participants assigned to the groups nor the evaluators who measure the variables know to which group the subjects belong.
  To be part of the study, participants must obtain high scores in anxiety (STAI questionnaire).
  The calculation estimates a sample of 36 participants: 18 for the experimental group and 18 for the placebo group.
  Participants will be randomly assigned to the experimental group or the placebo group.
  In addition to anxiety levels before and after treatment, variables such as chronic pain, central sensitization, general health, somatization and depression will be measured.
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be assigned to two groups:
  * Experimental group: who will receive myofascial intervention
  * Control / placebo group: who will receive sham myofascial intervention
  Neither the participants assigned to the groups nor the evaluators who measure the variables know to which group the subjects belong.
  Participants will be randomly assigned through the GraphPad software.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial treatment (Experimental): 4 sessions of myofascial intervention, 40 minutes per session, 1 session per week
  Interventions: Other: Myofascial treatment
- Sham myofascial treatment (Sham Comparator): 4 sessions of sham myofascial intervention, 40 minutes per session, 1 session per week
  Interventions: Other: Sham myofascial treatment

INTERVENTIONS:
Other: Myofascial treatment — 40 minutes of myofascial intervention: 10 min in each of the following regions with the patient face up:
  * Thoracolumbar fascia and abdomen
  * C7-T4 and sternum
  * Suboccipital area
  * Temporary area
  Arms: Myofascial treatment
Other: Sham myofascial treatment — 40 minutes of sham myofascial intervention: 10 min in each of the following regions with the patient face up and with the contact of the physiotherapist through a towel and without any intention:
  * Thoracolumbar fascia and abdomen
  * C7-T4 and sternum
  * Suboccipital area
  * Temporary area
  Arms: Sham myofascial treatment

SUMMARY:
This study evaluates the efficacy of a myofascial intervention as a technique within manual therapy in the treatment of clinical anxiety in adults. Half of the participants will receive a myofascial intervention program, while the other half will receive a sham myofascial intervention.

DETAILED DESCRIPTION:
Within physiotherapy, some studies have been carried out with psychological outcome measures, mainly from therapeutic exercise, but there continues to be an important documentary gap and the few results are not conclusive.

The myofascial approach is presented as an effective tool for the treatment of different pathologies, mainly musculoskeletal. However, few are the studies that relate it to psychological variables and specifically to improve anxiety levels.

The myofascial approach is proposed as a fast and low-cost tool for the management of clinical anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 and 65 years old
* Subjects with high levels of anxiety
* Subjects who speak and understand Spanish correctly
* Subjects without previous experience in myofascial treatment

Exclusion Criteria:

* Subjects with a clinical history of cognitive impairment
* Subjects with systemic, neurological or muscular diseases
* Subjects with some type of aneurysm diagnosed
* Subjects with diagnosed extremely high blood pressure
* Subjects with diagnosed malignant tumors
* Subjects with diagnosed vertebrobasilar insufficiency
* Subjects with a diagnosed dermatological condition
* Subjects diagnosed with epilepsy
* Pregnant women or with the possibility that they may be

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2022-07-29 (Actual)

PRIMARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | Change from baseline (pre-treatment), immediately after myofascial intervention (intrasession), through study completion (an average of 1 month), 3 and 6 months follow-up
  It consists of a self-report to evaluate two independent concepts about anxiety: anxiety as a state ("in this moment") and anxiety as a trait ("in most cases"). Each of these subscales has a total of 20 items in a 4-point Likert response system according to intensity (0 = not at all; 3 = a lot). The total score in each of the subscales ranges from 0 to 60 points.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | Change from baseline (pre-treatment), immediately after myofascial intervention (intrasession), through study completion (an average of 1 month), 3 and 6 months follow-up
  It consists of a horizontal line of 10 centimeters, at the ends of which appear "no pain" and "maximum pain". Patients mark where they would locate their intensity of chronic pain and later it is measured with a ruler indicating its result in millimeters.
Central Sensitization Inventory (CSI) | Change from baseline (pre-treatment), through study completion (an average of 1 month), 3 and 6 months follow-up
  Self-report to identify symptoms related to a central sensitization. It consists of a total of 25 items in a 5-point response system according to intensity (0 = never; 4 = always). The total score ranges from 0 to 100.
General Health Questionnaire (GHQ-12) | Change from baseline (pre-treatment), through study completion (an average of 1 month), 3 and 6 months follow-up
  Questionnaire to evaluate general health. It consists of a total of 12 items (6 of them positive sentences and 6 negative sentences) in a 4-point response system according to intensity (0-3). The total score ranges from 0 to 36.
Patient Health Questionnaire (PHQ-15) | Change from baseline (pre-treatment), through study completion (an average of 1 month), 3 and 6 months follow-up
  Questionnaire to evaluate somatic symptoms. It consists of a total of 15 items in a 2-point response system according to intensity (0 = not at all; 2 = a lot). The total score ranges from 0 to 30.
Beck Depression Inventory (BDI) | Change from baseline (pre-treatment), through study completion (an average of 1 month), 3 and 6 months follow-up
  Self-report to evaluate depressive symptoms. It consists of a total of 21 items in a 3-point response system according to intensity (0 = not at all; 3 = a lot). The total score ranges from 0 to 63.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Gozalo Pascual, PT, Principal Investigator — Universidad Complutense de Madrid
Locations (1):
- Pulsion Fisioterapia, Madrid, Spain

REFERENCES:
- [Derived] Gozalo-Pascual R, Gonzalez-Ordi H, Atin-Arratibel MA, Llames-Sanchez J, Alvarez-Melcon AC. Efficacy of the myofascial approach as a manual therapy technique in patients with clinical anxiety: A randomized controlled clinical trial. Complement Ther Clin Pract. 2023 May;51:101753. doi: 10.1016/j.ctcp.2023.101753. Epub 2023 Mar 29. PMID 37004342